CLINICAL TRIAL: NCT01132157
Title: The Comparison of Preconditioning Effect of Desflurane and Antiapoptotic Effect of Propofol in Patients With Kidney Transplantation
Brief Title: Comparison of the Protective Effect of Desflurane and Propofol in Patients With Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4-2009-0598
Record Dates: First submitted 2010-05-24; First posted 2010-05-27 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Healthy; End Stage Renal Disease
Keywords: Healthy Kidney Donors and Their Recipients with End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Desflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol group (Experimental)
  Interventions: Drug: Propofol
- Desflurane group (Active Comparator)
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Desflurane — In Desflurane group, donors and their recipients will be anesthetized with desflurane and remifentanil. In contrast, in Propofol group, donors will be anesthetized with Propofol and remifentanil and recipients will be anesthetized with desflurane and remifentanil.
  Arms: Desflurane group
Drug: Propofol — In Desflurane group, donors and their recipients will be anesthetized with desflurane and remifentanil. In contrast, in Propofol group, donors will be anesthetized with Propofol and remifentanil and recipients will be anesthetized with desflurane and remifentanil.
  Arms: Propofol group

SUMMARY:
Ischemia/reperfusion (IR) injury is the major cause of early renal dysfunction and acute renal failure of the transplanted kidney after renal transplantation. In 1986, Murry et al. described the phenomenon "ischemic preconditioning". Also, it was reported that a few non-ischemic stimuli could provide cellular tolerance against major ischemia through a mechanism similar to ischemic preconditioning. In an animal study, 1 minimal alveolar concentration of volatile anesthetics - a clinically relevant concentration - was reported to have a protective effect against ischemia/reperfusion injury, the effect being variable between types of anesthetics. Also, there were somm reports that intravenous anesthetics such as propofol could reduce IR injury by decreasing oxidative stress and apoptosis.

By reducing the ischemia/reperfusion injury of the grafted kidney, the morbidity and mortality related to renal transplantation can be reduced as well. The objective of this study is to find out whether, according to the type of anesthetics (Desflurane vs. Propofol), there is a difference in the protective effect against ischemia/reperfusion injury of the grafted kidney in patients receiving renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

* healthy kidney donors and their recipients of renal transplantation.

Exclusion Criteria:

* a donor that has any medical or surgical history,
* a recipient that is scheduled to have any other surgery with renal transplantation surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
BUN(Blood Urea Nitrogen) | 1 hour after surgery
  The primary outcome of our study is to find out whether, according to donors' anesthetics (desflurane or propofol), there is a difference in grafted kidney function postoperatively.
Cr density | 1 hour after surgery
  The primary outcome of our study is to find out whether, according to donors' anesthetics (desflurane or propofol), there is a difference in grafted kidney function postoperatively.
estimated GFR(Glomerular Filtration Ratio) | 1 hour after surgery
  The primary outcome of our study is to find out whether, according to donors' anesthetics (desflurane or propofol), there is a difference in grafted kidney function postoperatively.
urine output to check the the degree of protection for renal function | 1 hour after surgery
  The primary outcome of our study is to find out whether, according to donors' anesthetics (desflurane or propofol), there is a difference in grafted kidney function postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Bon Nyeo Koo, MD, Ph.D, Principal Investigator — Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Severance hospital, Yonsei University College of Medicine, Seoul, South Korea